CLINICAL TRIAL: NCT04149535
Title: PROTECTED TAVR: Stroke PROTECTion With SEntinel During Transcatheter
Brief Title: PROTECTED TAVR: Stroke PROTECTion With SEntinel During Transcatheter Aortic Valve Replacement
Acronym: PROTECTED TAVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2453
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Results first posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TAVR with Sentinel (Experimental): Patients assigned to this group will undergo TAVR with the Sentinel® Cerebral Protection System.
  Interventions: Device: Sentinel® Cerebral Protection System
- TAVR without Sentinel (No Intervention): Patients assigned to this group will undergo TAVR without the Sentinel® Cerebral Protection System.

INTERVENTIONS:
Device: Sentinel® Cerebral Protection System — cerebral embolic protection system
  Arms: TAVR with Sentinel

SUMMARY:
To demonstrate that use of the Sentinel® Cerebral Protection System significantly reduces the risk of peri-procedural stroke (≤72 hours) after transcatheter aortic valve replacement (TAVR).

ELIGIBILITY:
Inclusion Criteria:

* Subject has documented aortic valve stenosis and is treated with an approved TAVR device via transfemoral access
* Subject has the recommended artery diameter at the site of filter placement per the Sentinel® Cerebral Protection System Instructions For Use: 9-15 mm for the brachiocephalic artery and 6.5-10 mm in the left common carotid artery.
* Subject (or legal representative) provides written informed consent.

Exclusion Criteria:

* Subject has arterial stenosis >70% in either the left common carotid artery or the brachiocephalic artery.
* Subject's brachiocephalic or left carotid artery reveals significant stenosis, ectasia, dissection, or aneurysm at the aortic ostium or within 3 cm of the aortic ostium.
* Subject has compromised blood flow to the right upper extremity.
* Subject has access vessels with excessive tortuosity.
* Subject has uncorrected bleeding disorders.
* Subject is contraindicated for anticoagulant and antiplatelet therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir Kapadia, MD, Principal Investigator — The Cleveland Clinic
Locations (56):
- United States (41):
  - Tucson Medical Center, Tucson, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California, Davis Medical Center, Sacramento, California
  - Kaiser Foundation Hospital - San Francisco, San Francisco, California
  - Los Robles Regional Medical Center, Thousand Oaks, California
  - South Denver Cardiology Associates PC and Swedish medical center, Littleton, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Intercoastal Medical Group, Sarasota, Florida
  - Tampa General Hospital, Tampa, Florida
  - Piedmont Hosptial, Atlanta, Georgia
  - Wellstar, Marietta, Georgia
  - St. Johns Hospital, Springfield, Illinois
  - Community Munster, Munster, Indiana
  - Mercy Hospital Medical Center, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Lahey Clinic Hospital, Burlington, Massachusetts
  - Sparrow Hospital, Lansing, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Research Medical Center, Kansas City, Missouri
  - Creighton - Bergan Cardiology, Omaha, Nebraska
  - Englewood Medical Center, Englewood, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Kaleida Health, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - NYU Winthrop, Mineola, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Lankenau, Wynnewood, Pennsylvania
  - Baptist Memorial, Memphis, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - Vanderbilt, Nashville, Tennessee
  - Heart Hospital of Austin, Austin, Texas
  - Baylor Heart and Vascular, Dallas, Texas
  - The Methodist Hospital, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Baylor Scott and White, Round Rock, Texas
  - Methodist Healthcare System of San Antonio dba Methodist Hospital, San Antonio, Texas
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Australia (2):
  - Monash Medical Center, Clayton, Victoria
  - The Prince Charles Hospital, Chermside
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
- France (2):
  - CHU La Timone Hospital, Marseille
  - Clinique Pasteur, Toulouse
- Germany (6):
  - Heart Center Leipzig, Bad Segeberg
  - Herzzentrum Dresden GmbH, Dresden
  - University Hospital Frankfurt, Frankfurt
  - Universitaetsklinikum Schleswig-Holstein, Lübeck
  - LMU Klinikum der Universität München, Münich
  - Universitaetsklinikum Ulm, Ulm
- Italy (3):
  - Policlinico San Donato, San Donato, Milanese
  - Maria Cecilia Hospital SPA, Cotignola
  - Fondazione Centro San Raffaele, Milan

IPD SHARING:
Plan to Share IPD: Undecided
The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy (http://www.bostonscientific.com/en-US/data-sharing-requests.html)

REFERENCES:
- [Derived] Makkar RR, Gupta A, Waggoner TE, Horr S, Karha J, Satler L, Stoler RC, Alvarez J, Sakhuja R, MacDonald L, Modolo R, Leon MB, Linke A, Kapadia SR. Cerebral Embolic Protection by Geographic Region: A Post Hoc Analysis of the PROTECTED TAVR Randomized Clinical Trial. JAMA Cardiol. 2025 Jan 1;10(1):17-24. doi: 10.1001/jamacardio.2024.4278. PMID 39471309
- [Derived] Kapadia SR, Makkar R, Leon M, Abdel-Wahab M, Waggoner T, Massberg S, Rottbauer W, Horr S, Sondergaard L, Karha J, Gooley R, Satler L, Stoler RC, Messe SR, Baron SJ, Seeger J, Kodali S, Krishnaswamy A, Thourani VH, Harrington K, Pocock S, Modolo R, Allocco DJ, Meredith IT, Linke A; PROTECTED TAVR Investigators. Cerebral Embolic Protection during Transcatheter Aortic-Valve Replacement. N Engl J Med. 2022 Oct 6;387(14):1253-1263. doi: 10.1056/NEJMoa2204961. Epub 2022 Sep 17. PMID 36121045

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAVR With Sentinel | TAVR Without Sentinel
Started | 1501 | 1499
Completed | 1472 | 1481
Not Completed | 29 | 18
Not completed — Death | 11 | 7
Not completed — Physician Decision | 10 | 4
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Not described | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAVR With Sentinel | TAVR Without Sentinel | Total
Number analyzed (Participants) | 1501 | 1499 | 3000
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.9 (8.0) | 78.9 (7.8) | 78.9 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 631 | 566 | 1197
  Male | 870 | 933 | 1803
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Data not collected on patients from EU.
  Participants
    American Indian or Alaska Native: number analyzed (Participants) | 961 | 963 | 1924
    American Indian or Alaska Native | 5 | 3 | 8
    Asian: number analyzed (Participants) | 961 | 963 | 1924
    Asian | 14 | 16 | 30
    Black or African Heritage: number analyzed (Participants) | 961 | 963 | 1924
    Black or African Heritage | 31 | 25 | 56
    Caucasian: number analyzed (Participants) | 961 | 963 | 1924
    Caucasian | 852 | 872 | 1724
    Hispanic or Latino: number analyzed (Participants) | 961 | 963 | 1924
    Hispanic or Latino | 53 | 35 | 88
    Native Hawaiian or Other Pacific Islander: number analyzed (Participants) | 961 | 963 | 1924
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Other: number analyzed (Participants) | 961 | 963 | 1924
    Other | 12 | 13 | 25
    Not Disclosed: number analyzed (Participants) | 961 | 963 | 1924
    Not Disclosed | 11 | 11 | 22
Surgical Risk (Per Heart Team): Extreme/High Risk [Count of Participants; unit: Participants] — Risk of Mortality based on site specific Heart Team evaluation. There is not a defined scale.
  Participants | 457 | 456 | 913
Surgical Risk (Per Heart Team): Intermediate Risk [Count of Participants; unit: Participants] — Risk of Mortality based on site specific Heart Team evaluation. There is not a defined scale.
  Participants | 499 | 512 | 1011
Surgical Risk (Per Heart Team): Low Risk [Count of Participants; unit: Participants] — Risk of Mortality based on site specific Heart Team evaluation. There is not a defined scale.
  Participants | 545 | 531 | 1076
Native/Non-Native Valve Calcification Severity (site reported): None/Mild [Count of Participants; unit: Participants] | 241 | 223 | 464
Native/Non-Native Valve Calcification Severity (site reported): Moderate [Count of Participants; unit: Participants] | 418 | 426 | 844
Native/Non-Native Calcification Severity (site reported): Severe/Extreme [Count of Participants; unit: Participants] | 773 | 792 | 1565

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Stroke Through 72 Hours Post TAVR Procedure or Discharge (Whichever Comes First)
Description: All stroke (hemorrhagic, ischemic, or undetermined status; disabling or nondisabling) through 72 hours post TAVR procedure or discharge (whichever comes first), as adjudicated by an independent Clinical Events Committee (CEC) and using Neurologic Academic Research Consortium (NeuroARC) definitions.
Time Frame: <=72 hours
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | TAVR With Sentinel | TAVR Without Sentinel
Number analyzed (Participants) | 1501 | 1499
Participants | 34 | 43

ADVERSE EVENTS:
Time Frame: Events were reported to BSC from the time of enrollment through 72 hours or subject discharge (whichever comes first) for all patients. For patients with stroke within 72hrs/discharge, events were reported to BSC from the time of enrollment through 30+/-7 days post stroke. All-Cause Mortality includes all patients through 72 hours or subject discharge (whichever comes first), plus mortality through 30+/-7 days for patients that had stroke.
Description: All SAE, ADE, SADE, UADE, USADE, device deficiencies, and CEC events were reported to BSC.
Arm/Group | TAVR With Sentinel | TAVR Without Sentinel
All-Cause Mortality (participants affected / at risk) | 11/1501 | 7/1499
Serious Adverse Events (participants affected / at risk) | 285/1501 | 315/1499
Other Adverse Events (participants affected / at risk) | 0/1501 | 0/1499
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAVR With Sentinel (N=1501) | TAVR Without Sentinel (N=1499)
Atrioventricular block complete (Cardiac disorders) | 86 | 92
Bundle branch block left (Cardiac disorders) | 41 | 29
Atrial fibrillation (Cardiac disorders) | 15 | 14
Pericardial effusion (Cardiac disorders) | 8 | 6
Atrioventricular block second degree (Cardiac disorders) | 7 | 6
Atrioventricular block first degree (Cardiac disorders) | 6 | 6
Bradycardia (Cardiac disorders) | 5 | 7
Cardiac arrest (Cardiac disorders) | 8 | 3
Atrioventricular block (Cardiac disorders) | 4 | 5
Cardiac tamponade (Cardiac disorders) | 6 | 3
Cardiogenic shock (Cardiac disorders) | 5 | 4
Cardiac failure (Cardiac disorders) | 5 | 3
Ventricular tachycardia (Cardiac disorders) | 2 | 6
Bundle branch block right (Cardiac disorders) | 4 | 2
Aortic valve incompetence (Cardiac disorders) | 3 | 2
Ventricular fibrillation (Cardiac disorders) | 4 | 1
Bradyarrhythmia (Cardiac disorders) | 1 | 3
Cardiac failure congestive (Cardiac disorders) | 2 | 2
Mitral valve incompetence (Cardiac disorders) | 3 | 1
Sinus node dysfunction (Cardiac disorders) | 3 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Coronary artery occlusion (Cardiac disorders) | 2 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 1
Nodal arrhythmia (Cardiac disorders) | 1 | 1
Nodal rhythm (Cardiac disorders) | 2 | 0
Pericardial haemorrhage (Cardiac disorders) | 1 | 1
Prosthetic cardiac valve thrombosis (Cardiac disorders) | 1 | 1
Right ventricular failure (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 1
Bundle branch block (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1
Chronic left ventricular failure (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Coronary artery insufficiency (Cardiac disorders) | 0 | 1
Defect conduction intraventricular (Cardiac disorders) | 1 | 0
Myocardial haemorrhage (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial rupture (Cardiac disorders) | 0 | 1
Pulseless electrical activity (Cardiac disorders) | 1 | 0
Right ventricular dysfunction (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Torsade de pointes (Cardiac disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 9 | 18
Ischaemic stroke (Nervous system disorders) | 9 | 13
Transient ischaemic attack (Nervous system disorders) | 3 | 4
Cerebral infarction (Nervous system disorders) | 5 | 1
Embolic stroke (Nervous system disorders) | 2 | 1
Cerebral haemorrhage (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 1 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebellar stroke (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Lacunar infarction (Nervous system disorders) | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Vascular procedure complication (Injury, poisoning and procedural complications) | 9 | 15
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 6 | 11
Postoperative delirium (Injury, poisoning and procedural complications) | 2 | 2
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 3
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 2 | 1
Aortic annulus rupture (Injury, poisoning and procedural complications) | 1 | 1
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 1 | 1
Aortic pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 | 0
Device deployment issue (Injury, poisoning and procedural complications) | 1 | 0
Femoral nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Iatrogenic injury (Injury, poisoning and procedural complications) | 0 | 1
Post procedural fever (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 | 0
Hypotension (Vascular disorders) | 6 | 8
Arterial haemorrhage (Vascular disorders) | 4 | 3
Peripheral artery occlusion (Vascular disorders) | 2 | 4
Peripheral artery stenosis (Vascular disorders) | 3 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 4
Shock haemorrhagic (Vascular disorders) | 1 | 2
Aortic aneurysm (Vascular disorders) | 2 | 0
Aortic intramural haematoma (Vascular disorders) | 1 | 1
Aortic rupture (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0
Hypertensive emergency (Vascular disorders) | 1 | 1
Iliac artery occlusion (Vascular disorders) | 0 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 1
Shock (Vascular disorders) | 1 | 1
Aortic arteriosclerosis (Vascular disorders) | 1 | 0
Arteriovenous fistula (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Haemodynamic instability (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypertensive urgency (Vascular disorders) | 1 | 0
Hypoperfusion (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
Catheter site haemorrhage (General disorders) | 8 | 6
Pyrexia (General disorders) | 2 | 4
Catheter site haematoma (General disorders) | 1 | 4
Device embolisation (General disorders) | 3 | 1
Multiple organ dysfunction syndrome (General disorders) | 2 | 2
Calcinosis (General disorders) | 0 | 1
Extravasation (General disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 12 | 10
Haematuria (Renal and urinary disorders) | 2 | 2
Urinary retention (Renal and urinary disorders) | 1 | 2
Renal failure (Renal and urinary disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 7 | 6
Blood loss anaemia (Blood and lymphatic system disorders) | 4 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 10 | 10
Mental status changes (Psychiatric disorders) | 1 | 1
Device dislocation (Product Issues) | 3 | 3
Device failure (Product Issues) | 3 | 2
Device leakage (Product Issues) | 0 | 2
Device malfunction (Product Issues) | 2 | 0
Lead dislodgement (Product Issues) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 2
Corona virus infection (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 0 | 2
Infection (Infections and infestations) | 0 | 1
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Cardiovascular function test abnormal (Investigations) | 0 | 1
Electrocardiogram QRS complex prolonged (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Retinal artery occlusion (Eye disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/35/NCT04149535/Prot_SAP_000.pdf